CLINICAL TRIAL: NCT00872963
Title: An Extended Follow up of a Phase 2b Vaccine Trial With RTS,S/AS01E in Kilifi District, Kenya.
Brief Title: An Extended Follow up of a RTS,S/AS01E Malaria Vaccine Trial
Acronym: MAL059
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SSC 1512
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Malaria
Keywords: malaria vaccine; RTS,S,
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Yearly cross sectional bleeds to collect blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RABIES VACCINE: Those subjects who received the active comparator
  Interventions: Biological: RTS,S/AS01E
- RTS,S/AS01E: The subjects who received investigational product
  Interventions: Biological: RTS,S/AS01E

INTERVENTIONS:
Biological: RTS,S/AS01E — 0.5MLS of RTS,S/AS01E at 0,1,2 monthly schedule 0.5mls Rabies vaccine at 0,1,2 monthly schedule
  Other Names: rabies vaccine BP, Sanofi-Pasteur

SUMMARY:
Malaria is one of the leading causes of deaths in children below five years old. Despite antimalarial drugs and insecticide treated bed nets, the established means of treatment and protection, malaria still continues to affect many children. A malaria vaccine would be a very effective way of reducing malaria infection in the community. RTS,S/AS01E is a leading malaria vaccine candidate which is being developed for children in Africa. The investigators have done a study to find out if this vaccine is effective in reducing infection by malaria in children aged 5-17 months living in Kenya and Tanzania. The follow up of the original study was 14-18 months. The extended follow up is proposed to continue for another four years.

DETAILED DESCRIPTION:
The RTS,S/AS01E candidate malaria vaccine is being developed for the routine immunization of infants and children living in malaria-endemic areas as part of the Expanded Program of Immunization (EPI). 30% efficacy against clinical malaria and 58% efficacy against severe malaria disease was seen with a related vaccine, RTS,S/AS02A, in children aged 1 to 4 years (Malaria-026) in Mozambique. The efficacy against clinical malaria and infection was sustained beyond 18 months. The RTS,S/AS01 vaccines have been developed in parallel with the RTS,S/AS02 vaccines, and differ in the adjuvant formulation which has been shown to be more immunogenic.The utility of a partially effective vaccination depends heavily on the overall effect of malaria incidence during a child"s acquisition of natural immunity. However, other cohorts vaccinated in Phase II studies have already discontinued follow up for episodes of malaria, and the planned Phase III studies will run for at most 30 months post vaccination. The proposed extended follow up is expected to run for four years and will inform the design of Phase 4 studies and may prove critical in informing public health policy once the vaccine is licensed.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment and vaccination in the RTS,S/AS01E clinical trial (NCT00380393)
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child.

Exclusion Criteria:

* Moving out of the study area, so that follow up is impractical.

Ages: 19 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The local population is predominantly from Mijikenda ethnic group. The study area is within Kilifi District at the Kenyan coast and majority are subsistence farmers.Kilifi District experiences long rains in May-July and short rains in November/December. Measured Entomological Inoculation Rates in the area vary from 10-50 per year.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2009-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Long term febrile malaria episodes | 4 years

SECONDARY OUTCOMES:
To compare the age distribution of episodes of malaria following vaccination with RTS,S with the age distribution following control vaccination. | 4 years
To compare the in vitro markers of naturally acquired immunity in vaccinated and unvaccinated children, and assess the associations of these markers with subsequent episodes of febrile malaria. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ally Olotu, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (1):
- Kemri Wellcome Trust Research Programme, Kilifi, Coast Province, Kenya

REFERENCES:
- [Derived] Olotu A, Fegan G, Wambua J, Nyangweso G, Leach A, Lievens M, Kaslow DC, Njuguna P, Marsh K, Bejon P. Seven-Year Efficacy of RTS,S/AS01 Malaria Vaccine among Young African Children. N Engl J Med. 2016 Jun 30;374(26):2519-29. doi: 10.1056/NEJMoa1515257. PMID 27355532
- [Derived] Olotu A, Fegan G, Wambua J, Nyangweso G, Awuondo KO, Leach A, Lievens M, Leboulleux D, Njuguna P, Peshu N, Marsh K, Bejon P. Four-year efficacy of RTS,S/AS01E and its interaction with malaria exposure. N Engl J Med. 2013 Mar 21;368(12):1111-20. doi: 10.1056/NEJMoa1207564. PMID 23514288